CLINICAL TRIAL: NCT03479567
Title: Fine and Gross Motor Function and Relationship With Muscle Tone in Older Adults With and Without Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EC/2014/1240
Record Dates: First submitted 2018-03-13; First posted 2018-03-27 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Dementia; Gait; Balance; Muscle Tone; Fine Motor Function; Paratonia
MeSH Terms: conditions — Dementia; Muscle Rigidity

STUDY DESIGN:
Intervention Model Description: cross-sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HC (Other): Healthy controls, i.e. older adults without cognitive impairment
  Interventions: Other: Gait accelerometry; Other: balance accelerometry; Other: Fine motor skill test; Diagnostic Test: Paratonia Assessment Instrument (PAI); Other: myotonometric measurement of muscle tone
- MiD (Other): older adults with mild dementia
  Interventions: Other: Gait accelerometry; Other: balance accelerometry; Other: Fine motor skill test; Diagnostic Test: Paratonia Assessment Instrument (PAI); Other: myotonometric measurement of muscle tone
- MoD (Other): older adults with moderate dementia
  Interventions: Other: Gait accelerometry; Other: balance accelerometry; Other: Fine motor skill test; Other: myotonometric measurement of muscle tone

INTERVENTIONS:
Other: Gait accelerometry — accelerometric assessment of gait (Dynaport Hybrid): 7m walk in 3 conditions (normal pace, fast, double task)
Other: balance accelerometry — accelerometric assessment of balance (Dynaport Hybrid) during 10 seconds trial in 3 conditions (side-by-side, semitandem, tandem)
Other: Fine motor skill test — assessment of fine motor skills with Purdue Pegboard, with dominant hand, non-dominant hand and bimanual
Diagnostic Test: Paratonia Assessment Instrument (PAI) — diagnosis of paratonia based on passive movement of the four limbs
  Arms: HC; MiD
Other: myotonometric measurement of muscle tone — MyotonPRO measurement of muscle tone

SUMMARY:
The purpose of this study was (1) to investigate changes in gait, balance, fine motor function, and muscle tone, and (2) to find out if there is a correlation between muscle tone/presence of paratonia and motor function (gross and fine) in mild and moderate dementia.Three groups of participants were included in the study: healthy elderly (n=60), participants with mild dementia (n=31) and participants with moderate dementia (n=31). Measurements of fine motor function, balance, gait, presence of paratonia and muscle tone measurements were performed.

ELIGIBILITY:
Inclusion Criteria:

* age >= 65 years
* walk independently for at least 11 meters
* HC: no cognitive deterioration, MiD: dementia, Global Deterioration Scale<5, MoD: dementia, Global Deterioration Scale 5 or 6

Exclusion Criteria:

* recent (≤ 6 months) orthopedic surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 122 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
walking speed | through study completion, an average of 3 years
  gait speed parameter
step regularity | through study completion, an average of 3 years
  gait parameter representing regularity, autocorrelation (method Moe-Nilssen 2004), value between 0 and 1, with 1 representing perfect regularity
mediolateral jerk | through study completion, an average of 3 years
  balance smoothness and coordination, lower jerk values correspond with better smoothness of balance
anteroposterior jerk | through study completion, an average of 3 years
  balance smoothness and coordination, lower jerk values correspond with better smoothness of balance
Fine motor function | through study completion, an average of 3 years
  score on the Purdue pegboard test, maximal amount of (pairs of) pegs placed in 30 seconds (max. 25)
presence of paratonia | through study completion, an average of 3 years
  Paratonia Assessment Instrument, resistance against passive movements of the four limbs is evaluated (Hobbelen 2008)
MyotonPRO measurement of muscle tone | through study completion, an average of 3 years
  MyotonPRO measurement

SECONDARY OUTCOMES:
MyotonPRO measurement of elasticity | through study completion, an average of 3 years
  MyotonPRO measurement
MyotonPRO measurement of mechanical stiffness | through study completion, an average of 3 years
  MyotonPRO measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Vakgroep Revaki - Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided